CLINICAL TRIAL: NCT02751892
Title: Feasibility of a Physical Activity Intervention Informed by Self-Determination Theory With Patients Recovering From Colorectal Cancer
Brief Title: The Feasibility of an Active Lifestyle Programme in Patients Recovering From Colorectal Cancer
Acronym: MOVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of East Anglia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 13/EE/0060
Record Dates: First submitted 2016-04-21; First posted 2016-04-26 (Estimated); Last update posted 2016-04-26 (Estimated); Status verified 2016-04

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active Lifestyle Programme (Experimental): Supervised exercises for 3 months and motivational interviewing to facilitate physical activity behaviour change. Supervised exercise sessions took place twice per week for the first four weeks. This was tapered off to once per week for the second four weeks. During the last month of the intervention participants continued with the exercise at home and were encouraged to achieve 150min of moderate to vigorous PA per week.
  Interventions: Behavioral: Active lifestyle programme
- Standard Care (No Intervention): Received usual care. Was offered the intervention after the completion of the study.

INTERVENTIONS:
Behavioral: Active lifestyle programme — The intervention is an activity lifestyle programme to increase physical activity behaviour post-intervention and to facilitate behaviour change maintenance at 3 months post-intervention.
  Other Names: MOVE
  Arms: Active Lifestyle Programme

SUMMARY:
Long-term maintenance of physical activity behaviour change post-intervention remains challenging. This study is investigating the feasibility of a behaviour change intervention based on Self-Determination Theory in people recovering from colorectal cancer and its effects on behaviour change 6 months post-intervention.

DETAILED DESCRIPTION:
This study was a randomized controlled feasibility trial consisting of a 3-months active lifestyle intervention and a 3-months follow-up period. Participants were allocated to an active lifestyle programme (ALP) or the standard (SC) care group. ALP was offered 12 supervised exercise sessions over 3 months and six supportive behaviour change workshops. SC was encouraged to continue with their usual lifestyle. The intervention was informed by Self-Determination Theory.

The supervised exercise sessions took place in small groups of maximum 7 participants and lasted approximately 1 hour. Exercise included aerobic and resistance exercises. The behaviour change workshops were delivered in a motivational interviewing style, also in small groups of maximum 7 participants.

Participants were followed-up at 6 months. There was no contact with participants during the post-intervention and follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* a histologically confirmed diagnosis of colorectal cancer with Dukes stages A-C
* completed cancer treatment within the last 24 months,
* be able to understand spoken and written English
* score of 80 or more on the Karnofsky Performance Status Scale

Exclusion Criteria:

* already meeting general PA guidelines of 150 min of moderate PA or 75 min of vigorous intensity PA per week,
* recent myocardial infarction
* uncontrolled hypertension
* a pacemaker
* or unstable angina.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2013-10; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Change in minutes spent in moderate and vigorous intensity physical activity measure with the International Physical Activity Questionnaire long version | 0, 3, 6 months

SECONDARY OUTCOMES:
Change in behavioural regulation measure with the Behavioural Regulation in Exercise Questionnaire version 2 | 0, 3, 6 months
Change in psychological needs satisfaction measured with the psychological needs satisfaction in exercise scale | 0, 3, 6 months
Change in quality of life measure with the Functional Assessment of Cancer Therapy general | 0, 3, 6 months
Change in quality of life measure with the Functional Assessment of Cancer Therapy-colorectal | 0, 3, 6 months
Change in fatigue with the Functional Assessment of Cancer Therapy - fatigue | 0, 3, 6 months
Change in intention to exercise | 0, 3, 6 months
  assessed with Intention to exercise scale
Change in barriers to exercise | 0, 3, 6 months
  assessed with Barriers to Exercise scale
Change in physical fitness | 0, 3, and 6 months
  assessed with the modified Bruce treadmill test
Change in upper body strength-grip strength | 0, 3, 6 months
  Assessed with grip dynanometer
Change in upper body strength-upper arm strength | 0, 3, 6 months
  Assessed with biceps curl test
Change in lower body strength | 0, 3, 6 months
  Assessed with 30 sec sit-to-stand test
Changes in body composition (% body fat) assessed with bioelectrical impedance analysis | 0, 3, 6 months
Change in antropometric measures (waist circumference, hip circumference | 0, 3, 6 months
  Waist and hip circumference will be used to calculate the waist-to-hip ratio
Changes in anthropometric measures (height, weight, BMI) | 0, 3, 6 months
  Body weight and body height will be used to calculate BMI
Change in minutes spent in moderate and vigorous intensity physical activity with accelerometry | 0, 3, 6 months

CONTACTS AND LOCATIONS:
Overall Officials: John M Saxton, PhD, Principal Investigator — Northumbria University, Newcastle, United Kingdom

IPD SHARING:
Plan to Share IPD: No